CLINICAL TRIAL: NCT06082193
Title: Olfactory Cleft Stenosis and Obstruction on Paranasal Sinus CT Scan in Pre Septo Rhinoplasty Patients Without Respiratory Mucosa Pathology : Normal Variants or Pathologic Findings ?
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, JANKOWSKI Roger, Professor, Central Hospital, Nancy, France
Other Study IDs: 2023PI023
Record Dates: First submitted 2023-10-08; First posted 2023-10-13 (Actual); Last update posted 2023-10-13 (Actual); Status verified 2023-10

CONDITIONS: Olfactory Impairment
Keywords: Olfactory Cleft stenosis; Sniffin stick test; Non mucosa pathology; Olfactory recess; Olfactory Cleft Obstruction; Olfactory normal variant
MeSH Terms: conditions — Olfaction Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This retrospective studed included patients referred to our institution between December 2013 and december 2021 for septoplasty or septorhinoplasty. All patients underwent pre operatory paranasal sinus CT scan and olfactory test. Olfacory cleft stenosis will be quoted as none (less than 1/3 contact between nasal septum and ethmoïd turbinates), partial (1/3-2/3 contact between nasal septum and turbinates) or total (more than 2/3 contact between nasal septum and turbinates), as well as Olfactory Cleft obstruction as none (opacification less than 1/3 of olfactory cleft), partial (1/3-2/3 opacification) or complete (more than 2/3 opacification).

DETAILED DESCRIPTION:
In this retrospective study, We will include every patients over 18 years old who had a septoplasty or septorhinoplasty between December 2013 and December 2021 and who underwent paranasal CT scan and olfactory test (sniffin stick test).

The patients will be find thanks to social security code GAMA007 for septoplastie, GAMA 004, 010 for septorhinoplasty and olfactometry GJQP001.

The patients with mucosa pathology on CT scan or with record of chronic respiratory rhinitis, septum perforation or a pathology that can alter the olfaction on the consultation report will be excluded.

Olfactory measurements were performed before surgery using the threshold and identification subtests of Sniffin Stick Test. Olfactory status will be classified by taking into account the normative data provided by Hummel et al and the real identification score. The patients will be classified as normosmic if the threshold and the identification score is superior the tenth percentile. If not, they will be classified as anosmic if both score are 0 and hyposmic otherwise.

2 experienced radiologists will perform the measures on paranasal sinus CT. They will be blinded to olfactory results.

The olfactory cleft boundaries were determined in the coronal plane : Anterior boundary was defined by the anterior attachment of the middle turbinate; the posterior boundary corresponding to the anterior face of the sphenoid sinus; the lateral boundaries were defined as the attachment of the middle and/or superior turbinate laterally and the nasal septum medially. Olfactory clefts were divided into an anterior and a posterior compartment, defined as "middle olfactory recess" and "superior olfactory recess", laterally bounded by the middle and the superior turbinate lamella, respectively.

Each olfactory recess width, global olfactory Cleft width and cribriform plate width will be measured in the coronal plane, at the level of the cribriform plate and 5mm underneath at 5 different sites :

1. - First slice depicting the cribriform plate (entry of the middle olfactory recess)
2. - Middle of the middle olfactory recess (halfway throuh 1 and 3)
3. - First slice depicting the head of the superior turbinate (entry of the superior olfactory recess)
4. - Middle of the superior olfactory recess (halfway through 3 and 5)
5. - Anterior face of sphenoid sinus Olfactory cleft length will be determined in the sagittal plane as length of the cribriform plate.

Olfacory cleft stenosis will be quoted as none (less than 1/3 contact between nasal septum and ethmoïd turbinates), partial (1/3-2/3 contact between nasal septum and turbinates) or total (more than 2/3 contact between nasal septum and turbinates), A global olfactory cleft status will be obtained : no significant or partial stenosis in any compartment, total stenosis in case of complete stenosis in every compartment and intermediate stenosis in any other situation.

Olfactory Cleft obstruction will be classified as none (opacification less than 1/3 of olfactory cleft), partial (1/3-2/3 opacification) or complete (more than 2/3 opacification).

Olfactory cleft lateral boundaries will be evaluated for the presence of a lamellar pneumatization (superior, middle or lamellar concha bullosa).

Olfactory groove depth was classified according to the Keros classification in regard of the middle and superior olfactory recess.

as well as Olfactory Cleft obstruction as none (opacification less than 1/3 of olfactory cleft), partial (1/3-2/3 opacification) or complete (more than 2/3 opacification).

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years old who underwent paranasal sinus CT and olfactory test before septoplasty or septorhinoplasty

Exclusion Criteria:

* Respiratory mucosa pathology on CT (polyposis, opacification of the maxillary sinuses, ethmoid cells, frontal sinus, sphenoidal sinus, sinonasal tumor)
* septal perforation
* chronic respiratory rhinitis (allergic, vasomotor, mucoviscidosis)
* pathologie that can alter olfaction (multiple sclerosis, meningioma, post infection such as COVID)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: - Patients over 18 years old who underwent paranasal sinus CT and olfactory test before septoplasty or septorhinoplasty without respiratory mucosa pathology Sex, mean age Olfactory test threshold and identification using sniffin stick test. Classification normosmic or hyposmic using Hummel table.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2023-10-08 (Estimated); Study Completion 2023-10-25 (Estimated)

PRIMARY OUTCOMES:
Olfactory cleft stenosis or obstruction | 1 day
  Measures will classify as none, partial or total stenosis or obstruction

SECONDARY OUTCOMES:
Impact of olfactory cleft stenosis or obstruction | 1 day
  Are patients with stenosis or obstruction hypsomic or anosmic

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Jankowski Roger, Nancy
  - Centre Hospitalier Régional Universitaire - Service ORL, Nancy

IPD SHARING:
Plan to Share IPD: Undecided
The initial database of patients with olfactory measure and septoplasty or septorhinoplasty can be used for other research as well the one with the patients included (without mucosa pathology)

REFERENCES:
- [Background] Jafek BW, Murrow B, Michaels R, Restrepo D, Linschoten M. Biopsies of human olfactory epithelium. Chem Senses. 2002 Sep;27(7):623-8. doi: 10.1093/chemse/27.7.623. PMID 12200342
- [Background] Leboucq N, Menjot de Champfleur N, Menjot de Champfleur S, Bonafe A. The olfactory system. Diagn Interv Imaging. 2013 Oct;94(10):985-91. doi: 10.1016/j.diii.2013.06.006. Epub 2013 Aug 7. PMID 23932763
- [Background] Biacabe B, Faulcon P, Amanou L, Bonfils P. Olfactory cleft disease: an analysis of 13 cases. Otolaryngol Head Neck Surg. 2004 Feb;130(2):202-8. doi: 10.1016/j.otohns.2003.09.002. PMID 14990917
- [Background] Jankowski R, Rumeau C, Gallet P, Nguyen DT, Russel A, Toussaint B. Endoscopic surgery of the olfactory cleft. Eur Ann Otorhinolaryngol Head Neck Dis. 2018 Apr;135(2):137-141. doi: 10.1016/j.anorl.2017.09.005. Epub 2017 Oct 23. PMID 29074286
- [Background] Jankowski R, Nguyen DT, Gallet P, Rumeau C. Olfactory cleft dilatation. Eur Ann Otorhinolaryngol Head Neck Dis. 2018 Dec;135(6):437-441. doi: 10.1016/j.anorl.2018.05.008. Epub 2018 Jun 20. PMID 29934261
- [Background] Jiang RS, Liang KL. The Effect of Endoscopic Olfactory Cleft Opening on Obstructed Olfactory Cleft Disease. Int J Otolaryngol. 2020 Mar 27;2020:8073726. doi: 10.1155/2020/8073726. eCollection 2020. PMID 32292482
- [Background] Kuperan AB, Lieberman SM, Jourdy DN, Al-Bar MH, Goldstein BJ, Casiano RR. The effect of endoscopic olfactory cleft polyp removal on olfaction. Am J Rhinol Allergy. 2015 Jul-Aug;29(4):309-13. doi: 10.2500/ajra.2015.29.4191. PMID 26163252
- [Background] Nguyen DT, Bey A, Arous F, Nguyen-Thi PL, Felix-Ravelo M, Jankowski R. Can surgeons predict the olfactory outcomes after endoscopic surgery for nasal polyposis? Laryngoscope. 2015 Jul;125(7):1535-40. doi: 10.1002/lary.25223. Epub 2015 Mar 5. PMID 25752823
- [Background] Nguyen DT, Gauchotte G, Nguyen-Thi PL, Jankowski R. Does surgery of the olfactory clefts modify the sense of smell? Am J Rhinol Allergy. 2013 Jul-Aug;27(4):317-21. doi: 10.2500/ajra.2013.27.3907. PMID 23883814
- [Background] Chang H, Lee HJ, Mo JH, Lee CH, Kim JW. Clinical implication of the olfactory cleft in patients with chronic rhinosinusitis and olfactory loss. Arch Otolaryngol Head Neck Surg. 2009 Oct;135(10):988-92. doi: 10.1001/archoto.2009.140. PMID 19841336
- [Background] Kohli P, Schlosser RJ, Storck K, Soler ZM. Olfactory cleft computed tomography analysis and olfaction in chronic rhinosinusitis. Am J Rhinol Allergy. 2016 Nov 1;30(6):402-406. doi: 10.2500/ajra.2016.30.4365. PMID 28124650
- [Background] Loftus C, Schlosser RJ, Smith TL, Alt JA, Ramakrishnan VR, Mattos JL, Mappus E, Storck K, Yoo F, Soler ZM. Olfactory cleft and sinus opacification differentially impact olfaction in chronic rhinosinusitis. Laryngoscope. 2020 Oct;130(10):2311-2318. doi: 10.1002/lary.28332. Epub 2019 Oct 11. PMID 31603563
- [Background] Soler ZM, Pallanch JF, Sansoni ER, Jones CS, Lawrence LA, Schlosser RJ, Mace JC, Smith TL. Volumetric computed tomography analysis of the olfactory cleft in patients with chronic rhinosinusitis. Int Forum Allergy Rhinol. 2015 Sep;5(9):846-54. doi: 10.1002/alr.21552. Epub 2015 May 26. PMID 26010298
- [Background] Eliezer M, Hamel AL, Houdart E, Herman P, Housset J, Jourdaine C, Eloit C, Verillaud B, Hautefort C. Loss of smell in patients with COVID-19: MRI data reveal a transient edema of the olfactory clefts. Neurology. 2020 Dec 8;95(23):e3145-e3152. doi: 10.1212/WNL.0000000000010806. Epub 2020 Sep 11. PMID 32917809
- [Background] Altundag A, Yildirim D, Tekcan Sanli DE, Cayonu M, Kandemirli SG, Sanli AN, Arici Duz O, Saatci O. Olfactory Cleft Measurements and COVID-19-Related Anosmia. Otolaryngol Head Neck Surg. 2021 Jun;164(6):1337-1344. doi: 10.1177/0194599820965920. Epub 2020 Oct 13. PMID 33045908
- [Background] Tekcan Sanli DE, Altundag A, Yildirim D, Kandemirli SG, Sanli AN. Comparison of Olfactory Cleft Width and Volumes in Patients with COVID-19 Anosmia and COVID-19 Cases Without Anosmia. ORL J Otorhinolaryngol Relat Spec. 2022;84(1):1-9. doi: 10.1159/000518672. Epub 2021 Sep 21. PMID 34569549
- [Background] Alves de Sousa F, Tarrio J, Sousa Machado A, Costa JR, Pinto C, Nobrega Pinto A, Moreira B, Meireles L. Olfactory Cleft Length: A Possible Risk Factor for Persistent Post-COVID-19 Olfactory Dysfunction. ORL J Otorhinolaryngol Relat Spec. 2023;85(3):119-127. doi: 10.1159/000527141. Epub 2022 Nov 1. PMID 36318894
- [Background] Lima NB, Jankowski R, Georgel T, Grignon B, Guillemin F, Vignaud JM. Respiratory adenomatoid hamartoma must be suspected on CT-scan enlargement of the olfactory clefts. Rhinology. 2006 Dec;44(4):264-9. PMID 17216743
- [Background] Kandemirli SG, Altundag A, Yildirim D, Tekcan Sanli DE, Saatci O. Olfactory Bulb MRI and Paranasal Sinus CT Findings in Persistent COVID-19 Anosmia. Acad Radiol. 2021 Jan;28(1):28-35. doi: 10.1016/j.acra.2020.10.006. Epub 2020 Oct 19. PMID 33132007
- [Background] Jankowski R, Rumeau C, Gallet P, Nguyen DT. Nasal polyposis (or chronic olfactory rhinitis). Eur Ann Otorhinolaryngol Head Neck Dis. 2018 Jun;135(3):191-196. doi: 10.1016/j.anorl.2018.03.004. Epub 2018 Apr 13. PMID 29661611
- [Background] Whyte A, Boeddinghaus R. Imaging of adult nasal obstruction. Clin Radiol. 2020 Sep;75(9):688-704. doi: 10.1016/j.crad.2019.07.027. Epub 2019 Sep 9. PMID 31515050
- [Background] Hummel T, Kobal G, Gudziol H, Mackay-Sim A. Normative data for the "Sniffin' Sticks" including tests of odor identification, odor discrimination, and olfactory thresholds: an upgrade based on a group of more than 3,000 subjects. Eur Arch Otorhinolaryngol. 2007 Mar;264(3):237-43. doi: 10.1007/s00405-006-0173-0. Epub 2006 Sep 23. PMID 17021776
- [Background] Nguyen DT, Rumeau C, Gallet P, Jankowski R. Olfactory exploration: State of the art. Eur Ann Otorhinolaryngol Head Neck Dis. 2016 Apr;133(2):113-8. doi: 10.1016/j.anorl.2015.08.038. Epub 2015 Sep 15. PMID 26384780